CLINICAL TRIAL: NCT02318524
Title: Circulation of Pathogenic Fungi in the Domestic Environment: Clinical Impact of Mould and Pneumocystis Jirovecii Exposure on COPD Patients
Brief Title: Clinical Impact of Fungal Domestic Environmental Exposure on COPD Patients
Acronym: FungiCOPD
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Région Nord-Pas de Calais, France (Other); Pfizer (Industry); Merck Sharp & Dohme LLC (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010_35; 2010-A01379-30 (Other: ID RCB number, ANSM)
Record Dates: First submitted 2013-04-22; First posted 2014-12-17 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: COPD; Pulmonary Fungal Diseases; Environmental Exposure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Fungal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum, serum, oropharyngeal washing, Dust catchers
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Fungal infections could play a role in chronic obstructive pulmonary disease (COPD) patient's exacerbations and in lung function impairment. In fact, Aspergillus fumigatus is often isolated from respiratory samples, but few data are available about its clinical significance. Aspergillus colonization could be associated to a higher risk of invasive pulmonary aspergillosis (IPA), which, in COPD patients, is characterized by a 2% incidence (probably underestimated) and a high mortality (72 to 95%). Similarly, detection of anti-Aspergillus antibodies is quite frequent in COPD patients but its significance and usefulness for aspergillosis diagnosis and follow-up have not been assessed. Furthermore, several studies suggest a frequent carriage of Pneumocystis jirovecii, reaching 37-55%, with a higher frequency in the most severe COPD stages and a possible role of colonisation in the occurrence and progression of COPD.

As these colonization and sensitization phenomena could be related to domestic exposure to airborne or, for P. jirovecii, to human reservoirs, the investigators set-up a study in order to (i) Evaluate how domestic exposure to mould or to P. jirovecii could impact fungal colonization and sensitization frequency in COPD patients, (ii) Study the relationship between these fungal colonization/sensitization phenomena and lung function impairment in the course of COPD and (iii) Have a better understanding of mould and P. jirovecii circulation in the close environment of patients (between airborne, human reservoirs and patients).

In fine, this study will provide data (i) On fungal contamination levels (species and conidia concentration) of COPD patient's homes in a French region, (ii) On the relationship between fungal exposure level and colonization/sensitization phenomena, (iii) On the role of fungal colonization/sensitization in lung function impairment, (iv) To design diagnostic, therapeutic, and preventive options for the management of COPD patients, taking into account fungal environmental exposure and colonization/sensitization impact on the evolution of the disease.

DETAILED DESCRIPTION:
The investigators will focus on both the patient and its domestic environment. More precisely, for 80 patients, the investigators will measure mould domestic exposure (determination of mould frequency during an environmental investigation at the patient's home), search for mould sensitization and colonization (complete bio clinical check-up including spirometry, inflammatory and mycological markers at inclusion), and do a clinical follow-up of exacerbation's (frequency and severity). At last, clinical and environmental mould and P. jirovecii isolates will be characterized at the phenotypic and genotypic level.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 90 years old male or female,
* COPD patient (I to IV stages),
* Medical consultation or severe COPD exacerbation requiring hospitalization.

Exclusion Criteria:

* Active tuberculosis.
* Cancer (or prior anticancer therapy within the past 3 years).
* Diffuse bronchiectasia.
* Cystic fibrosis.
* Asthma.
* Any other pulmonary disease (sarcoidosis, pulmonary fibrosis, pneumoconiosis,…).
* Prior anti- P. jirovecii or antifungal treatment within the past 6 months.
* Pregnant or breast-feeding females.
* Patient with no social insurance.
* Patient unwilling to comply with the protocol.
* Patient unable to understand the study and its objectives.
* Patient under guardianship.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2011-08; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Comparison of domestic mould exposure of colonized/sensitized and non colonized/non sensitized COPD patients. | Mould exposure and colonization/sensitization will be measured at inclusion. Patients will undergo a bioclinical checkup 18 months after inclusion.
  The primary endpoint will be the difference between " colonized/sensitized " and " non colonized/non sensitized " groups in change of mould exposure level. Mould exposure level is a numeric value which corresponds to the concentration of fungal conidia in the dust catcher (measurement by culture and quantitative real-time PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Fréalle, PharmD, PhD, Study Director — Lille University Hospital; Stéphanie Fry, MD, Principal Investigator — Lille University Hospital
Locations (1):
- Lille University Hospital, Lille, France

IPD SHARING:
Plan to Share IPD: No